CLINICAL TRIAL: NCT05010226
Title: Focused Ultrasound for the Treatment of Pancreatic Cancer - an International Registry
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202007081RINB
Record Dates: First submitted 2021-07-27; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Pancreatic Cancer; Focused Ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the registry is to collect data on the performance of the focused ultrasound (FUS) technology and health outcomes. A wide variety of approaches exist for using FUS on pancreatic cancer patients, and the primary goal is to capture this broad spectrum of approaches and their impact on patients overall health. This information will help provide a better understanding of current care, and may possibly direct further, more specific investigations that will follow this registry.

DETAILED DESCRIPTION:
This is a single-group, multi-center, observational log-in study. Patients will be screened for clinically diagnosed pancreatic cancer and are scheduled to receive focused ultrasound therapy at National Taiwan University Hospital to determine their eligibility for participation. After confirming that the patient has agreed, the patient will be followed up for 12 months to observe safety, tumor response, changes in clinical manifestations, and changes in the process of focused ultrasound treatment and quality of life after treatment. The overall survival and disease progression time will be tracked within 3 days before and after the 7th day of focused ultrasound treatment to death or 12 months, with the earlier occurrence being the priority. The patient's survival status will be tracked for 1 year.

The physical condition will be evaluated by laboratory tests during the baseline screening, the next day after treatment, and 7 days, 14 days, 1 month, 2 months, 3 months, 6 months, and 12 months. Including blood tests, serum biochemical tests, tumor indicators, etc.; quality of life assessment, including pain index score (VAS) and SF-36 life scale (The MOS item short-form health survey, SF-36) will be one after treatment Evaluation starts in the following month; MRI imaging examination, all examinations, and treatments have been carried out in the 201701032DIPD clinical trial case. This case is only an observational clinical trial case for data registration.

The baseline screening before treatment will be carried out between the -3 days and the 0 days before the treatment. The overall survival time (OS) will be tracked for 1 year; the time to disease progression (TTP) and progression-free survival (PFS) will continue to be tracked during the trial until the patient dies or undergoes other curative procedures (tracking should be carried out every 3 months) once). Concomitant drugs/treatments and adverse events will be tracked continuously during the trial period.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this registry, an individual must meet all of the following criteria:

  1. 20 years and older
  2. Provision of signed and dated informed consent form
  3. Stated willingness to comply with all registry procedures and availability for the duration of the registry
  4. Histology proven pancreatic carcinoma in any area of pancreas
  5. Pancreatic tumor that can be treated by FUS
  6. Willingness and ability to complete follow-up interviews
  7. Patients have agreed to participate in the clinical trial 201701032DIPD and were scheduled to receive FUS therapy in our hospital

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this registry:

  1. Any disease, condition or surgery which would result in a contraindication to undergoing FUS therapy.
  2. Clinical trials of pancreatic cancer not of focused ultrasound or related activities

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will be implemented at approximately 10 sites internationally. In order to achieve the target registry population of 30 participants over 12 months in the NTUH site, participants who receive focused ultrasound for pancreatic cancer. Participant enrollment will be evaluated on a site by site basis throughout the enrollment period to provide diversity of participant and system representation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pain related to pancreatic cancer | after high focused ultrasound treatment, an average of 1 month
  Brief Pain Inventory from 0 (no pain) to 10 (pain as a bad as can imagine)
To observe the efficacy of local tumor ablation | after high focused ultrasound treatment, an average of 1 month
  the assessment of the tumor burden after high focused ultrasound treatment
The effect of local tumor ablation | over 12 months
  time-to-progression
To observe the survival rate | over 12 months
  overall survival (OS)
To observe the progression-free survival rate | over 12 months
  observation of the progression-free survival
To evaluate clinical benefit response (CBR) | over 12 months
  The proportion of participants with a CBR will be measured at each follow-up time point

OTHER OUTCOMES:
Impact on Quality of Life and Cost | over 12 months
  Standardized instrument to measure of health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, M.D. Ph.D, Principal Investigator — National Taiwan University Hospital